CLINICAL TRIAL: NCT00986011
Title: Effects of A Smart Growth Community on Prevention of Family Obesity Risks
Brief Title: Study of a Smart Growth Community's Effect on Prevention of Obesity in Middle-, Moderately Low- and Low-Income Families
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mary Ann Pentz, USC/Norris Comprehensive Cancer Center and Hospital
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: LAC-USC-HS-0700681; CDR0000655182 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-09-26; First posted 2009-09-29 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2009-09

CONDITIONS: Healthy, no Evidence of Disease; Obesity; Weight Changes
Keywords: obesity; weight changes; healthy, no evidence of disease
MeSH Terms: conditions — Obesity; Body Weight Changes

INTERVENTIONS:
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Other: survey administration
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Overweight and obesity have been associated with multiple types of disease, including cancer. Living in a smart growth community may encourage behaviors that would reduce the risk of obesity.

PURPOSE: This research study is looking at the effect of a smart growth community on prevention of obesity in middle-, moderately low- and low-income families.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effects of the whole set as well as individual smart growth principles on prevention of obesity risk in middle, moderately low, and low-income families who reside in a smart growth community, the Preserve, compared to two types of control groups of families who reside in other communities that may naturally vary in exposure to these principles.
* To evaluate the longitudinal-mediational relationship between increased activity and pro-health attitudes achieved in the smart growth community to lower obesity risk.
* To identify trajectories of physical activity over time and evaluate their relationship to obesity risk, including high-stable, early-onset stable, early-onset short-term, and low-stable trajectories.

Secondary (exploratory)

* To evaluate demographic x type of community (smart growth vs other) interactions (with the major ethnic groups representing Hispanic vs white), gender, parent vs child on outcomes, as well as on obesogenic trajectories.
* To evaluate a possible "chaining" or translational effect, i.e., whether effects of living in a smart growth community generalize to changes in eating behavior as part of a general change in health attitudes.
* To assess whether neighborhoods where physical activity actually takes place (defined as 0.5 square-mile area and 10-15 walking distance from residence, school [for children], work or equivalent [for index adult], and leisure), contribute significantly to physical activity and eating behavior beyond the effect of smart growth community residence.
* To determine whether some individual smart growth principles may have a relatively greater impact on obesity risk than others, in both intervention and control communities.
* To assess whether physical activity trajectories other than those hypothesized can be identified for their predictive relationship to obesity prevention.

OUTLINE: Participants receive an accelerometer monitor and are instructed to wear it for 7 continuous days (except when sleeping, bathing, or swimming) on the right hip attached to an adjusted belt to assess physical activity. Participants also undergo anthropometric measures (height and weight) using a calibrated digital scale and professional stadiometer.

Participants complete surveys and questionnaires on Self-reported Physical Activity, Self-reported Dietary Intake, and Social Network Survey. Participants also complete other self-reported items assessing demographic characteristics, family finances, health status, health history, length of current residence, home-relocation patterns, time use and transportation patterns, substance use, depression, sleeping habits, fast-food consumption, and school and work addresses.

PROJECTED ACCRUAL: A total of 390 families living in The Preserve, 195 families who were not chosen to live in The Preserve, and 195 control families who live in the surrounding area will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet 1 of the following criteria:

  * Residents who live in The Preserve, a smart growth community in Chino, California

    * Chosen by lottery to live in The Preserve
  * Prospective buyers and renters for residences in The Preserve (but were not chosen to live in The Preserve) living in the following communities and/or cities:

    * Ontario
    * Pomona
    * Diamond Bar
    * Corona
    * Yorba Linda/Mira Loma
    * Chino
  * Families from Chino and surrounding communities within a 30-minute drive from The Preserve
* Families with children in grades 4-8 must meet the following criteria:

  * Each family unit consists of 1 index parent defined as the parent who spends relatively more time in the neighborhood on a daily basis
  * An index child defined as a 4th-8th-grade child
* Income levels range from very-low income to middle income ($20-$165,000) based on Area Median Income

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2008-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Levels of physical activity and pro-healthy lifestyle attitudes
Body-mass index
Trajectories of physical activity and the relationship to obesity risk

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Pentz, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States

REFERENCES:
- [Derived] Dunton GF, Liao Y, Almanza E, Jerrett M, Spruijt-Metz D, Pentz MA. Locations of joint physical activity in parent-child pairs based on accelerometer and GPS monitoring. Ann Behav Med. 2013 Feb;45 Suppl 1(Suppl 1):S162-72. doi: 10.1007/s12160-012-9417-y. PMID 23011914